CLINICAL TRIAL: NCT03796143
Title: A Randomized Controlled Trial (RCT) Comparing Acceptance and Commitment Therapy (ACT) and Cognitive Behavioral Therapy (CBT) Self-help Books for Depression
Brief Title: Evaluation of Self-help Books for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Associate Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9766
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two active self-help interventions, or their choice of intervention, for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT self-help book condition (Experimental): Participants in this condition will be asked to read The Mindfulness and Acceptance Workbook for Depression by Strosahl and Robinson (2008), a self-help book based on acceptance and commitment therapy.
  Interventions: Behavioral: The Mindfulness and Acceptance Workbook for Depression
- CBT self-help book condition (Active Comparator): Participants in this condition will be asked to read Cognitive Behavioral Workbook for Depression by Knaus (2006), a self-help book based on acceptance and commitment therapy.
  Interventions: Behavioral: The Cognitive Behavioral Workbook for Depression
- Choice of two self-help books (Other): Participants in this condition will have the option of receiving either the self-help book by Strosahl and Robinson (2008) or the book by Knaus (2006).
  Interventions: Behavioral: The Mindfulness and Acceptance Workbook for Depression; Behavioral: The Cognitive Behavioral Workbook for Depression

INTERVENTIONS:
Behavioral: The Mindfulness and Acceptance Workbook for Depression — Participants assigned to this condition will be asked to read this self-help book over an 8-week period.
  Arms: ACT self-help book condition; Choice of two self-help books
Behavioral: The Cognitive Behavioral Workbook for Depression — Participants assigned to this condition will be asked to read this self-help book over an 8-week period.
  Arms: CBT self-help book condition; Choice of two self-help books

SUMMARY:
The goal of this study is to compare the efficacy of acceptance and commitment therapy (ACT) and cognitive behavioral therapy (CBT) for depression in a bibliotherapy format and assess hypothesized mechanisms of change in depression symptomatology, quality of life, and functioning.

This study will test the following hypotheses:

1. CBT and ACT will both result in decreased depression, distress, and self-stigma associated with depression. Life satisfaction and values progress will increase in both conditions.
2. CBT will result in greater use of reappraisal than ACT.
3. ACT will results in greater use of defusion and decreased psychological inflexibility than CBT.
4. Changes in experiential avoidance and defusion will predict changes in depression in the ACT condition.
5. Changes in reappraisal will predict changes in depression in the CBT condition.
6. Participants who are given their choice of treatment will show better adherence and satisfaction in the intervention.

DETAILED DESCRIPTION:
The investigators aim to recruit 150 participants for this RCT (50 per treatment condition). This will provided adequate power (0.80) to detect differences between groups of medium effect size (d=0.50). Note that detailed eligibility criteria are listed in the "Eligibility" section. Participants will be recruited via SONA, flyers, online postings, classroom announcements, and through the USU CBS lab website.

All study procedures will be completed online, on a computer/mobile phone. After completing informed consent online through Qualtrics, participants will complete an online baseline survey. Participants will then be randomized to one of three groups: a CBT book, an ACT book, or a choice between the two books. Participants will be asked not to access other self-help books during the study duration. A link will be provided to access the book online along with a 10-week suggested reading schedule. Participants will be asked to complete a midtreatment survey 5 weeks after the beginning of treatment, and a posttreatment survey 10 weeks after the beginning of treatment. A follow-up survey will be sent to participants 3 months after the posttreatment survey. In addition to psychological measures, these surveys will also ask about adherence and use of strategies taught in the book. Researcher contact will involve reminders to complete assessments and weekly reminders of the suggested reading schedule.

Participants assigned to the CBT condition will receive a link to access The Cognitive Behavioral Workbook for Depression (Knaus, 2008), based on a psychosocial treatment that has shown effectiveness in reducing depression symptoms (Jiménez, 2012). The primary treatment components in this book are psychoeducation (introducing the cognitive behavioral model of depression), self-assessment worksheets (e.g. identifying depressive thought patterns, separating sensations from appraisals), cognitive restructuring, using metacognition/logic, and avoiding perfectionism.

Participants assigned to the ACT condition will receive a link to access The Mindfulness and Acceptance Workbook for Depression (Strosahl & Robinson, 2008), based on a modern cognitive behavioral therapy that combines acceptance and mindfulness methods with values and behavior change methods (Hayes, Strosahl & Wilson, 2011). The primary treatment components in this book are psychoeducation (introducing the ACT model of depression), values and goals, mindfulness, acceptance, defusion, committed action, and "rewriting" inflexible life stories.

An additional subset of study participants will be given their choice of the two self-help books described above after completing the baseline assessment. Participants who are randomized to receive their choice of book will be provided a brief description of the contents of each book before making a decision.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Enrolled at Utah State University
* Have not participated in other self-help studies run by the USU CBS Lab
* Interested in using self-help book for depression
* Elevated depressive symptoms as determined by scoring a 10 or higher on the depression subscale of the Depression, Anxiety, and Stress Scale (DASS-21)

Exclusion Criteria:

* Below the age of 18
* Not a student at Utah State University
* Have participated in other self-help studies run by the USU CBS Lab
* Not interested in using self-help book for depression
* No elevated depressive symptoms as determined by scoring lower than 10 on the depression subscale of the Depression, Anxiety, and Stress Scale (DASS-21)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  Depression, Anxiety and Stress Scale (DASS) : a self-report measure of depression, anxiety, and stress symptoms. Higher scores indicate higher negative emotional states of depression, anxiety, and stress. This measure assesses each of these symptoms as a distinct subscale. Items are rated on a 4-point scale ranging from 0 "did not apply to me at all" to 3 "applied to me very much, or most of the time." Ranges for depression, anxiety, and stress are 0-28, 0-20, and 0-33, respectively.

SECONDARY OUTCOMES:
Self-Stigma of Depression Scale (SSDS; Barney, Griffiths, Christensen, & Jorm, 2010) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The SSDS is a 16-item measure of self-directed stigma about one's own experience of depression and consists of subscales of shame, self-blame, social inadequacy, and help-seeking inhibition. The measure generates four subscales for shame, self-blame, help-seeking inhibition, and feelings of social inadequacy, with higher scores indicating greater presence of these experiences. The subscales are summed to calculate a total score which ranges from 16 to 80, with higher scores indicating greater overall self-stigma.
Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The AAQ-II is a 10-item measure of psychological inflexibility and experiential avoidance. Items are rated on a 7-point scale ranging from 1 "never true" to 7 "always true." A total score is calculated by reverse coding so that higher scores indicate greater psychological flexibility.
Cognitive Fusion Questionnaire (CFQ; Gillanders et al., 2014) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The CFQ is a 7-item measure of cognitive fusion. Items are rated on a 7-point scale, ranging from 1 "never true" to 7 "always true." Total scores range from 7 to 49 with higher scores indicating greater levels of cognitive fusion.
The Behavioral Activation for Depression Scale (BADS; Kanter, Mulick, Busch, Berlin, & Martell, 2007) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The BADS is a 25-item measure of approach and avoidance behaviors in depression, separated into two subscales. Two additional subscales measure work/school and social impairment due to depressive symptoms. Within each subscale, higher scores indicate greater frequency of these behaviors.
Automatic Thoughts Questionnaire-Frequency (ATQ-30; Hollon & Kendall, 1980) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The ATQ is a 30-item measure of the frequency of automatic negative self-statements associated with depression. Items are rated on a 5-point scale, ranging from 1 "not at all" to 5 "all the time," with higher scores indicating a greater frequency of automatic thoughts.
Thought Control Questionnaire-Reappraisal Subscale (TCQ; Wells & Davies, 1994) | Baseline, midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline), and follow-up (3-months after posttreatment)
  The TCQ-Reappraisal subscale is 6-item measure of cognitive reappraisal of negative thoughts. Items are rated on a 4 point scale ranging from 1 "never" to 4 "almost always" indicating the frequency of cognitive reappraisal of negative thoughts. Total scores range from 6 to 24, with higher scores indicating greater frequency of cognitive reappraisal of negative thoughts.

OTHER OUTCOMES:
Adherence to self-help book | Midtreatment (5 weeks after baseline), posttreatment (10 weeks after baseline)
  Participants will be asked to rate their adherence to the exercises in the book with a single question on 7-point scale from "Did all recommended assignments" to "Did no recommended assignments," with higher scores indicating a greater proportion of the assignments were completed. This is adapted from previous studies of self-help adherence (Abramowitz, Moore, Braddock, & Harrington, 2009).
Satisfaction with self-help book | Posttreatment (10 weeks after baseline)
  Participants will be asked to rate 7 items evaluating their satisfaction with the self-help book on a 6-point scale from "Strongly disagree" to "Strongly agree." The scale produces a total score ranging from 7 to 42, with higher scores indicating greater satisfaction with the book. These items have been used to evaluate program satisfaction in previous self-help research conducted by our lab (e.g., Levin, Pierce, & Schoendorff, in press).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abramowitz JS, Moore EL, Braddock AE, Harrington DL. Self-help cognitive-behavioral therapy with minimal therapist contact for social phobia: a controlled trial. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):98-105. doi: 10.1016/j.jbtep.2008.04.004. Epub 2008 Apr 26. PMID 18514614
- [Background] Barney LJ, Griffiths KM, Christensen H, Jorm AF. The Self-Stigma of Depression Scale (SSDS): development and psychometric evaluation of a new instrument. Int J Methods Psychiatr Res. 2010 Dec;19(4):243-54. doi: 10.1002/mpr.325. PMID 20683846
- [Background] Beaufort IN, De Weert-Van Oene GH, Buwalda VAJ, de Leeuw JRJ, Goudriaan AE. The Depression, Anxiety and Stress Scale (DASS-21) as a Screener for Depression in Substance Use Disorder Inpatients: A Pilot Study. Eur Addict Res. 2017;23(5):260-268. doi: 10.1159/000485182. Epub 2017 Dec 8. PMID 29224000
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Fledderus M, Bohlmeijer ET, Pieterse ME, Schreurs KM. Acceptance and commitment therapy as guided self-help for psychological distress and positive mental health: a randomized controlled trial. Psychol Med. 2012 Mar;42(3):485-95. doi: 10.1017/S0033291711001206. Epub 2011 Jul 11. PMID 21740624
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K. G. (2011). Acceptance and commitment therapy: The process and practice of mindful change. Guilford Press.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Hollon, S. D., & Kendall, P. C. (1980). Cognitive self-statements in depression: Development of an automatic thoughts questionnaire. Cognitive Therapy and Research, 4(4), 383-395.
- [Background] Jiménez, F. J. R. (2012). Acceptance and commitment therapy versus traditional cognitive behavioral therapy: A systematic review and meta-analysis of current empirical evidence. International Journal of Psychology and Psychological Therapy, 12(3), 333-358.
- [Background] Fuhr K, Hautzinger M, Krisch K, Berking M, Ebert DD. Validation of the Behavioral Activation for Depression Scale (BADS)-Psychometric properties of the long and short form. Compr Psychiatry. 2016 Apr;66:209-18. doi: 10.1016/j.comppsych.2016.02.004. Epub 2016 Feb 9. PMID 26995255
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Knaus, W. J. (2006). The cognitive behavioral workbook for depression: a step-by-step program. New Harbinger Publications.
- [Background] Levin, M. E., Haeger, J., & Cruz, R. A. (2018). Tailoring Acceptance and Commitment Therapy Skill Coaching in the Moment Through Smartphones: Results from a Randomized Controlled Trial. Mindfulness, 1-11.
- [Background] Levin ME, Pistorello J, Seeley JR, Hayes SC. Feasibility of a prototype web-based acceptance and commitment therapy prevention program for college students. J Am Coll Health. 2014;62(1):20-30. doi: 10.1080/07448481.2013.843533. PMID 24313693
- [Background] Lorenzo-Luaces L, German RE, DeRubeis RJ. It's complicated: The relation between cognitive change procedures, cognitive change, and symptom change in cognitive therapy for depression. Clin Psychol Rev. 2015 Nov;41:3-15. doi: 10.1016/j.cpr.2014.12.003. Epub 2014 Dec 24. PMID 25595660
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Maslej MM, Bolker BM, Russell MJ, Eaton K, Durisko Z, Hollon SD, Swanson GM, Thomson JA Jr, Mulsant BH, Andrews PW. The Mortality and Myocardial Effects of Antidepressants Are Moderated by Preexisting Cardiovascular Disease: A Meta-Analysis. Psychother Psychosom. 2017;86(5):268-282. doi: 10.1159/000477940. Epub 2017 Sep 14. PMID 28903117
- [Background] Masuda, A., & Tully, E. C. (2012). The role of mindfulness and psychological flexibility in somatization, depression, anxiety, and general psychological distress in a nonclinical college sample. Journal of Evidence-Based Complementary & Alternative Medicine, 17(1), 66-71.
- [Background] Mohr DC, Hart SL, Howard I, Julian L, Vella L, Catledge C, Feldman MD. Barriers to psychotherapy among depressed and nondepressed primary care patients. Ann Behav Med. 2006 Dec;32(3):254-8. doi: 10.1207/s15324796abm3203_12. PMID 17107299
- [Background] Reynolds M, Wells A. The Thought Control Questionnaire--psychometric properties in a clinical sample, and relationships with PTSD and depression. Psychol Med. 1999 Sep;29(5):1089-99. doi: 10.1017/s003329179900104x. PMID 10576301
- [Background] Ridgway N, Williams C. Cognitive behavioural therapy self-help for depression: an overview. J Ment Health. 2011 Dec;20(6):593-603. doi: 10.3109/09638237.2011.613956. PMID 22126636
- [Background] Rokke PD, Tomhave JA, Jocic Z. The role of client choice and target selection in self-management therapy for depression in older adults. Psychol Aging. 1999 Mar;14(1):155-69. doi: 10.1037//0882-7974.14.1.155. PMID 10224639
- [Background] Strosahl, K. D., & Robinson, P. J. (2008). The mindfulness and acceptance workbook for depression: Using acceptance and commitment therapy to move through depression and create a life worth living. New Harbinger Publications.
- [Background] Tompkins KA, Swift JK, Callahan JL. Working with clients by incorporating their preferences. Psychotherapy (Chic). 2013 Sep;50(3):279-83. doi: 10.1037/a0032031. PMID 24000835
- [Background] van Schaik DJ, Klijn AF, van Hout HP, van Marwijk HW, Beekman AT, de Haan M, van Dyck R. Patients' preferences in the treatment of depressive disorder in primary care. Gen Hosp Psychiatry. 2004 May-Jun;26(3):184-9. doi: 10.1016/j.genhosppsych.2003.12.001. PMID 15121346
- [Background] Wells A, Davies MI. The Thought Control Questionnaire: a measure of individual differences in the control of unwanted thoughts. Behav Res Ther. 1994 Nov;32(8):871-8. doi: 10.1016/0005-7967(94)90168-6. PMID 7993332
- [Background] Wing RR, Phelan S, Tate D. The role of adherence in mediating the relationship between depression and health outcomes. J Psychosom Res. 2002 Oct;53(4):877-81. doi: 10.1016/s0022-3999(02)00315-x. PMID 12377297